CLINICAL TRIAL: NCT05417217
Title: The Effect of Continued Mechanical Ventilation on the Occurrence of Myocardial Ischemia in Patients Undergoing Totally Endoscopic Coronary Artery Bypass Grafting
Brief Title: The Effect of Continued Mechanical Ventilation on the Occurrence of Myocardial Ischemia
Acronym: VENTMICS-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the passing of the principal investigator, the clinical trial could not be continued.
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: f/2022/096
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Hypoxia
Keywords: Cardiac surgery; Minimally invasive cardiac surgery; Endoscopic coronary artery bypass grafting; Harlequin syndrome; Ventilation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Ischemia; Hypoxia; Harlequin syndrome; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Ventilation is discontinued after going on CPB and lungs are exposed to atmospheric pressure.
  Blood will be drawn:
  At baseline: before general anaesthesia, after start of CPB, after clamping the aorta, before unclamping the aorta, after the operation, 5 h after clamping the aorta, 12 hours after clamping the aorta, and 24 hours after aortic clamping
  Interventions: Procedure: Discontinued ventilation
- Ventilation group (Experimental): Ventilation is continued from going on CPB until clamping of the ascending aorta.
  Blood will be drawn:
  At baseline: before general anaesthesia, after start of CPB, after clamping the aorta, before unclamping the aorta, after the operation, 5 h after clamping the aorta, 12 hours after clamping the aorta, and 24 hours after aortic clamping
  Interventions: Procedure: Continued ventilation

INTERVENTIONS:
Procedure: Discontinued ventilation — Ventilation is discontinued after going on CPB and lungs are exposed to atmospheric pressure
  Arms: Control group
Procedure: Continued ventilation — Ventilation is continued from going on CPB until clamping of the ascending aorta with tidal volume 3ml/kg ideal body weight, Fraction of inspired oxygen (FiO2) 50%, respiratory rate 5/min and Inspiratory:Expiratory (I/E) ratio 1/2.
  Arms: Ventilation group

SUMMARY:
The goal of this study is to examine the influence of mechanical ventilation on the occurrence of myocardial ischemia in patients undergoing endo-CABG.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) surgery is one of the main treatment options for patients suffering from coronary artery disease, a condition characterized by a build-up of cholesterol in the coronary arteries of the heart that affects 126 million people worldwide each year. During this procedure, cardiopulmonary bypass (CPB) takes over the function of the heart and lungs. In recent years, there has been a huge focus on reducing surgical trauma in this procedure, leading to the emergence of minimally invasive cardiac surgery (MICS) such as endoscopic CABG (endo-CABG). In these techniques, peripheral CPB with femoral arterial cannulation is the most commonly used strategy. However, the use of retrograde arterial perfusion is not without risk. It can cause that the upper part of the body only receives deoxygenated blood. The effect on the heart is not yet fully known. The hypoxemia could cause myocardial ischemia and this could damage the heart muscle cells.

It is reported in the literature that establishing adequate ventilation from the initiation of CPB to cardiac arrest can resolve this phenomenon. This approach was investigated in a recently performed double-blinded, randomized, controlled pilot study (n=10) of our research group. However, a larger randomized controlled trial was needed. Therefore, this research aims to investigate the effect of continued mechanical ventilation on the occurrence of myocardial ischemia in patients undergoing endo-CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients undergoing their first elective endo-CABG procedure using peripheral cannulation for CPB
* Patients who are able to give their informed consent
* Patients who speak Dutch or French

Exclusion Criteria:

* Patients participating in another clinical trial
* Patients taking corticosteroids
* Patients with an ejection fraction < 25%
* Patients with lung diseases (chronic obstructive pulmonary disease (COPD), asthma)
* Patients where groin cannulation is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
The influence of continued mechanical ventilation on the release of cardiac troponin T (cTn-T) | Until 24 hours after clamping the aorta
  Cardiac troponin T is represented in ng/L. If the value of cTn-T exceeds 14 ng/L, then cTn-T is able to detect myocardial ischemia at the predefined time points.
The influence of continued mechanical ventilation on the release of creatine kinase-myocardial band (CK-MB) | Until 24 hours after clamping the aorta
  Creatine kinase-myocardial (CK-MB) band is represented in µg/L. If the value of CK-MB exceeds 6.2 µg/L, then CK-MB is able to detect myocardial ischemia at the predefined time points.
The influence of continued mechanical ventilation on the release of heart-type fatty acid-binding protein (hFABP) | Until 5 hours after clamping the aorta
  Heart-type fatty acid-binding protein (hFABP) is represented in ng/L. If the value of hFABP exceeds 6 ng/L, then hFABP is able to detect myocardial ischemia at the predefined time points.
The influence of continued mechanical ventilation on lipid peroxidation | Until unclamping the aorta (on average until 64 minutes after clamping the aorta)
  Lipid peroxidation is measured using the malondialdehyde assay.
The influence of continued mechanical ventilation on the redox balance | Until unclamping the aorta (on average until 64 minutes after clamping the aorta) ]
  superoxide dismutase 1 and 2 (SOD1, SOD2), nuclear factor erythroid 2-related factor 2 (Nrf2), catalase (CAT), glutathione peroxidase (GPx), NADPH oxidase 2 and 4 (NOX2, NOX4), heme oxygenase-1 (HO-1), NAD(P)H quinone oxidoreductase 1 (NQO-1)) will be studied to determine the redox balance.
The influence of continued mechanical ventilation on the partial pressure of oxygen (pO2) | Until the end of surgery (on average until 203 minutes after the start of the surgery)
  pO2 is represented in mmHg. If pO2 is lower than 60 mmHg, then hypoxemia is present.
The influence of continued mechanical ventilation on the partial pressure of carbon dioxide (pCO2) | Until the end of surgery (on average until 203 minutes after the start of the surgery)
  pCO2 is represented in mmHg.
The influence of continued mechanical ventilation on the pH | Until the end of surgery (on average until 203 minutes after the start of the surgery)
  The pH will measure the acidity.
The influence of continued mechanical ventilation on lactate | Until the end of surgery (on average until 203 minutes after the start of the surgery)
  Lactate is represented in mmol/L.

SECONDARY OUTCOMES:
The occurence of myocardial infarction | Until 30 days after surgery
  This is based on the Fourth universal definition of myocardial infarction (2018).
The occurence of mortality | Until 30 days after surgery
  All-cause mortality is evaluated.
The occurence of neurological complications | Until 30 days after surgery
  Neurological complications include cerebrovascular accident (CVA), transient ischemic attack (TIA), delirium, epilepsy
The occurence of graft failure | Until 30 days after surgery
  Graft failure describes total graft occlusion that prevents blood flow through the graft to the revascularized part of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Alaaddin Yilmaz, MD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No